CLINICAL TRIAL: NCT04819997
Title: A Nurse-Led Intervention for Fear of Progression in Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20594; NCI-2021-01138 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20594 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Lung Carcinoma; Metastatic Malignant Female Reproductive System Neoplasm; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (videoconference, questionnaire, survey) (Experimental): Patients participate in 5 videoconference sessions over 30 minutes each over 6 weeks focused on worry management skills, values-based goal setting, and brief mindfulness-based practices, then complete patient workbook activities after each session over 15-20 minutes per day. Patients also complete a survey over 8 minutes at 6 weeks, an exit interview at 7 weeks, and questionnaires over 25 minutes each at baseline, 6 weeks, and 10 weeks.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Participate in videoconference session
  Other Names: Education for Intervention

SUMMARY:
This clinical trial focuses on a nurse-led program that is designed to help patients cope with worries, fears, and uncertainty about the future. The purpose of this study is to understand if the program is helpful and practical to carry out at medical centers and community clinics. This study may help patients learn more effective ways to cope and respond to your concerns and any unhelpful thoughts.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and acceptability of the revised day by day (DBD) intervention in an academic and community settings.

II. To assess the preliminary effects of the revised DBD intervention for reducing fear of progression (FOP) and improving distress, anxiety, depression, metacognitions (beliefs about worry), and mindfulness.

OUTLINE:

Patients participate in 5 videoconference sessions over 30 minutes each over 6 weeks focused on worry management skills, values-based goal setting, and brief mindfulness-based practices, then complete patient workbook activities after each session over 15-20 minutes per day. Patients also complete a survey over 8 minutes at 6 weeks, an exit interview at 7 weeks, and questionnaires over 25 minutes each at baseline, 6 weeks, and 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III or IV gynecologic (GYN) or lung cancer
2. At least 3 months from initial diagnosis
3. Score >= 34 on the Fear of Progression-short form (SF) questionnaire

Exclusion Criteria:

1. Severe mental illness (e.g. psychosis)
2. Hospice enrolled
3. Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Up to 10 weeks
  Defined by enrollment rate. Enrollment rate will be calculated as number of enrolled divided by the number of eligible patients.
Feasibility of the intervention | Up to 10 weeks
  Defined by attrition, attendance, and adherence with home practice activities. Attrition rate will be calculated as number of patients who drop out patients divided by number of enrolled patients. Adherence will be assessed based on the completion rate of home practice activities.
Acceptability | Up to 10 weeks
  Will be assessed based on 1) responses to open-ended questions on the exit interview response asking about participants' experience with the intervention and delivery platforms; and 2) a self-report evaluation survey rating usefulness of the session content, home practice activities, testimonials, and delivery platforms. Survey items are rated on a 1-5 Likert scale. An average score of 3 or above will indicate good acceptability.

OTHER OUTCOMES:
Fear of progression (FOP) | Up to 10 weeks
  Linear mixed model (LMM) for repeated-measures design will be used to examine the changes in FOP and other outcome measures across three time-points. The model will include the time factor, employ compound symmetry covariance structure, and adjust for covariates when necessary. Post Hoc pairwise comparisons with Tukey adjustment will be conducted to test the change in outcomes between time periods. Cohen's D will be used to estimate effect sizes for the changes in outcome measures across time-points (Lakens, 2013).
Cancer-specific distress | Up to 10 weeks
  Cancer-specific distress assessed using the Impact of Event Scale-Revised (IES-R) [ Time Frame: Up to week 10 ] Cancer-specific distress will be assessed using the Impact of Event Scale-Revised (IES-R) , 22-item scale consisting of 3 subscales
  1. Intrusion;
  2. Avoidance; and
  3. Hyperarousal. Items are scored on a 0-4 response format. Subscale scores are calculated by taking the mean of the subscale responses. Total scores range from 0-88. A score of 24 or greater indicates clinical levels of distress.
Anxiety | Up to 10 weeks
  Anxiety will be assessed using the PROMIS-Anxiety 8a, measures fear, dread, worry, hyperarousal, and related somatic symptoms.
  The short-form consists of 8 items that are scored on a 0-5 response format. The raw score is calculated by summing the values of the response to each question (range 8-40).
  Scores are standardized such that the scale produces continuous T scores with a mean of 50 and a SD of 10, higher scores reflect higher distress.
  PROMIS T score thresholds for anxiety are: ˂ 55 normal; 55-64 mild; 65-74 moderate; ≥75 severe.
Depression | Up to 10 weeks
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9), includes the two major symptom domains: affective and somatic symptoms.
  It is rated from a 0 (not at all) to 3 (nearly every day) scale. Items are summed and a score of 10 or greater is considered clinically significant symptoms of depression.
  Scores of 0-4, 5-9, 10-14, and ≥15 represent minimal, mild, moderate, and severe levels of symptom burden.
Metacognitions | Up to 10 weeks
  Metacognitions (MCQ-30) will be assessed using the Metacognitions Questionnaire, MCQ-30 is a 30-item questionnaire that assesses beliefs about worry.
  It consists of 5 subscales: Positive beliefs about worry; Negative beliefs about worry, Cognitive confidence; Need to control thoughts; and Cognitive self-consciousness. For each subscale, items are scored 1-4 and subscale scores range from 6-24.
  Total scores range from 30 to 120; higher scores indicate more dysfunctional metacognitions.
Mindfulness | Up to 10 weeks
  Mindfulness will be assessed using the Five Facet Mindfulness Questionnaire (FFMQ-15), the FFMQ-15 assesses five facets of mindfulness: observing, describing, acting with awareness, non-reactivity, and non-judging of inner experience.
  Items are rated on a 5-point Likert scale ranging from 1 (never or rarely true) to 5 (very often or always true).
  3 items comprise each subscale and subscale scores range from 3-15. Higher scores indicate greater engagement with mindfulness skills.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reb, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States